CLINICAL TRIAL: NCT02194530
Title: Pilot Study to Collect Blood From Research Subjects Allergic and Non-allergic to Peanut to Study Immune Modulation With Anti-IgE Therapy in Mice
Brief Title: Reduction of Peanut Reactivity and Immune Modulation With Anti-IgE Therapy
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1405015102
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Peanut Allergy
Keywords: Peanut allergic individuals; Allergic/atopic individuals (not allergic to peanut); Non-allergic individuals
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Peanut allergic individuals: 20 individuals will be recruited for this group. Each blood draw will require 105 ml of whole blood to be collected in ten heparinized 10 mL tubes and one EDTA tube.
- Allergic/atopic individuals (not peanut): Subjects should not be allergic to peanut. 20 individuals will be recruited for this group. Each blood draw will require 105 ml of whole blood to be collected in ten heparinized 10 mL tubes and one EDTA tube.
- Non-allergic individuals: 20 individuals will be recruited for this group. Each blood draw will require 105 ml of whole blood to be collected in ten heparinized 10 mL tubes and one EDTA tube.

SUMMARY:
This pilot study is will examine the pathways involved in allergic response, primarily in food allergy; specifically peanut allergy. We will also study non-allergic donors as well as patients with atopic disorders, primarily as control subjects. We believe that this study will lead to discovery of significant pathways involved in the allergic pathway that can be explored in more detail during follow-up studies in order to address mechanistic questions that cannot be answered in a pilot trial. We believe that such a pilot study represents the ideal approach to identify effective therapeutic interventions and to simultaneously better understand the underlying mechanistic properties involved in the allergy cascade. We think that this study forms the basis for a novel avenue of research into the pathogenesis of allergic pathways, a disease that is still associated with significant morbidity and mortality.

DETAILED DESCRIPTION:
The study aims to characterize the pathways involved in the allergic response, primarily in food allergy; specifically peanut allergy. We will also study non-allergic donors as well as patients with atopic disorders, primarily as control subjects. All eligible study participants will have documented elevated total IgE levels, peanut positivity or another antigen/allergen specific elevated IgE (ie common indoor/outdoor allergens) prior to being enrolled in the study. Our study will focus on allergic as well as non-allergic individuals. We plan on collecting samples from a total of 60 patients during one time point (peanut allergic individuals, non-atopic/allergic individuals, atopic individuals-other than peanut allergy). We believe that such a pilot study represents the ideal approach to identify effective therapeutic interventions and to simultaneously better understand the underlying mechanistic properties involved in the allergy cascade. We plan to obtain a detailed history prior to enrollment as well as objective data (ie SPT as well as Immunocap testing results). There will be 3 study groups and studies will be performed on approximately 20 peanut allergic patients, 20 non-allergic controls, and 20 allergic/atopic (non-peanut allergic, but allergic to indoor/outdoor allergen) individuals. There will be one blood draw required at each visit (weeks 0, 4, 8). Each blood draw will require 105 ml of whole blood to be collected in ten heparinized 10-mL tubes and one EDTA tube. We plan to assess the levels of total IgE and IgG as well as antigen specific IgG and IgE in the peripheral blood of patients. We will specifically perform ELISA testing that detects these levels. We will also perform in vitro CD4+ T cell proliferation assays. For this purpose, patients' peripheral T cells will be isolated with a combination of magnetic beads and flow cytometric sorting.

ELIGIBILITY:
Inclusion Criteria for Groups 1-3:

Group 1: Peanut allergic individuals (n=20)

* 18-65 years of age
* Positive ImmunoCAP test (Optional)
* Documented elevated total IgE levels, peanut positivity or another antigen/allergen specific elevated IgE (ie common indoor/outdoor allergens)
* Experienced at least one of the following symptoms within 60 minutes of exposure:

  * Skin-related symptom (i.e., hives and edema)
  * Respiratory-related symptom (i.e., wheezing, throat tightness, repetitive coughing, and dyspnea)
  * Gastrointestinal-related symptom (i.e., vomiting and diarrhea)

Group 2: Allergic/atopic individuals (not allergic to peanut; n=20)

* 18-65 years of age.
* Positive ImmunoCAP test (Optional)
* Documented elevated total IgE levels or an indoor/outdoor antigen/allergen (other than peanut) specific elevated IgE (ie common indoor/outdoor allergens).
* Experienced at least one of the following symptoms within 60 minutes of exposure:

  * Skin-related symptom (i.e., hives and edema).
  * Respiratory-related symptom (i.e., wheezing, throat tightness, repetitive coughing, and dyspnea).
  * Gastrointestinal-related symptom (i.e., vomiting and diarrhea)

Group 3: Non-allergic individuals (healthy controls; n=20)

* 18-65 years of age.
* Negative ImmunoCAP test (Optional)
* Documented absence or low total IgE levels, or negativity for an antigen/allergen specific elevated IgE (ie common indoor/outdoor allergens).
* Has not experienced at least one of the following symptoms within 60 minutes of exposure to a particular substance:

  * Skin-related symptom (i.e., hives and edema).
  * Respiratory-related symptom (i.e., wheezing, throat tightness, repetitive coughing, and dyspnea).
  * Gastrointestinal-related symptom (i.e., vomiting and diarrhea)

Exclusion Criteria for Groups 1-3:

* Prior therapy with anti-IgE
* Steroid use greater than 10 mg/d prednisone or equivalent 30 days prior to enrollment
* Any immunosuppressive drug use within 3 months prior to screening (mycophenolate mofetil, hydroxychloroquine, azathioprine, methotrexate, leflunomide, rituximab, cyclophosphamide, intravenous immunoglobulin, plasmapheresis)
* Ongoing chronic infection (viral, bacterial or fungal) including known HIV, Hepatitis B/C
* Acute infection receiving any antibiotics within 30 days prior to screening
* Probiotics (greater than estimated 109 cfu or organisms per day) within 30 days prior to enrollment (with the exception of fermented beverages, milks or yogurts).
* Malignancy within one year prior to screening (with the exception of non-metastatic squamous or basal cell skin carcinomas and cervical carcinoma if received curative surgical treatment)
* Known illicit drug or alcohol abuse
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New York Metropolitan area residents
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2016-07-19 (Actual); Study Completion 2016-07-19 (Actual)

PRIMARY OUTCOMES:
Blood test to determine peanut allergy and peanut specific IgE and IgG | 1 year
  There will be one blood draw at each visit (weeks 0, 4, 8). Each blood draw will require 105 mL of whole blood to be collected in ten heparinized 10 mL tubes and one EDTA tube. We plan to assess the levels of total IgE and IgG as well as antigen specific IgG and IgE in the peripheral blood of patients. We will specifically perform ELISA testing that detects these levels. We will also perform in vitro CD4+ T cell proliferation assays.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Cornell Medical College, NY
Locations (1):
- Department of Genetic Medicine, Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided